CLINICAL TRIAL: NCT04042194
Title: Comparison of Connective Tissue Graft (CTG) and Titanium Prepared Platelet-Rich Fibrin (T-PRF) Inserted With a Double Layer Technique on Peri-Implant Soft Tissue Thickening: A Randomized Prospective Clinical Study
Brief Title: Comparison of CTG and T-PRF on Peri-Implant Soft Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Gulbahar, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018/68
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Peri-implant Mucositis; Peri-Implantitis; Thin Gingiva
Keywords: clinical research; Implant; Implantology; Prospective; Randomized controlled trial; Soft Tissue Grafting; Single-Tooth Implants
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thickened with T-PRF (Experimental): Following local anaesthesia, the measurement of soft tissue thickness at three points [1) occlusal part of the alveolar crest (OAC), 2) midbuccal mucosa level (MBML), 3) over 1 mm of mucogingival junction (MGJ1)] was performed with an endodontic spreader and digital caliber. Following the mid-crestal incision, the buccal flap was raised with double layer technique, while the lingual flap was left to enable direct visibility. The implant bed was drilled according to the manufacturer's protocol. The implants (BEGO Semados® RS/RSX implant system, Bremen, Germany) were placed at the bony crest. Right after the implant placement, the randomisation procedure was performed. In this group, the implants were placed in thin tissues, and T-PRF was inserted in the prepared mucoperiosteal flap at the facial site and secured with horizontal mattresses.
  Interventions: Procedure: Placement of Implants and Thickening Peri-Implant Mucosa with T-PRF
- Thickened with CTG (Active Comparator): Following local anaesthesia, the measurement of soft tissue thickness at three points [1) occlusal part of the alveolar crest (OAC), 2) midbuccal mucosa level (MBML), 3) over 1 mm of mucogingival junction (MGJ1)] was performed with an endodontic spreader and digital caliber. Following the mid-crestal incision, the buccal flap was raised with double layer technique, while the lingual flap was left to enable direct visibility. The implant bed was drilled according to the manufacturer's protocol. The implants (BEGO Semados® RS/RSX implant system, Bremen, Germany) were placed at the bony crest. Right after the implant placement, the randomisation procedure was performed. In this group, the implants were placed in thin tissues, and CTG was inserted in the prepared mucoperiosteal flap at the facial site and secured with horizontal mattresses.
  Interventions: Procedure: Placement of Implants and Thickening Peri-Implant Mucosa with CTG

INTERVENTIONS:
Procedure: Placement of Implants and Thickening Peri-Implant Mucosa with T-PRF — A total of 40 ml blood sample was collected from the antecubital vein of the patients' right or left arms with 10 ml injectors. 40 ml blood was transferred to a grade-IV titanium tube for the T-PRF group. The titanium tubes containing the blood samples were instantly centrifuged in a tabletop centrifuge at room temperature. The blood samples of the T-PRF group were centrifuged clockwise at 2700 RPM for 20 minutes. Subsequent to the centrifugation process, the clots of the T-PRF group were removed from the tubes with sterile tweezers, separated from the RBC base with scissors, and left for over 20 minutes on sterile woven gauze to release the serum slowly from the collected clots. The implants were placed in thin tissues, and the thickness of the thin tissues was simultaneously increased with T-PRF.
  Arms: Thickened with T-PRF
Procedure: Placement of Implants and Thickening Peri-Implant Mucosa with CTG — The implants were placed in thin tissues, and the thickness of the thin tissues was simultaneously increased with CTG. Autogenous connective tissue graft was harvested according to a single incision technique.
  Arms: Thickened with CTG

SUMMARY:
The present study aimed to increase the thickness of the gingiva and prevent possible crestal bone resorption by placing the CTG or T-PRF membrane under the mucosa immediately after the implant treatment in individuals with thin gingival phenotype. The null hypothesis was that T-PRF used simultaneously with implant placement can be considered an alternative to CTG.

DETAILED DESCRIPTION:
Although connective tissue graft (CTG) is considered as the best technique for soft tissue augmentation, limited supply of donor tissue because of palatal vessels and nerves, and postoperative pain may require alternative methods.

The purpose of this study is to reduce the crestal bone resorption around the implant site by augmenting the Peri-Implant Soft Tissue with T-PRF (titanium prepared platelet-rich fibrin) or CTG and to compare the effectiveness of the two techniques.

Through simultaneous augmentation of the soft tissue by T-PRF or CTG, a total of 30 implants were implanted in 30 patients (12 males, 18 females) with a mean age of 38.4 years. In the test group, implants were placed in thin tissues and thickened with T- PRF membrane at the same time, while in the control group, implants were placed in thin tissues and thickened with CTG at the same time. During the surgery (T 0 ) and at postoperative 3 months (T 1 ), keratinised tissue width (KTW) and Peri-Implant soft tissue thickness (STT) were measured from three points: occlusal part of the alveolar crest (OAC), midbuccal mucosa level (MBML), and over 1 mm of mucogingival junction (MGJ1).

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years,
* thin gingiva biotype,
* one missing tooth in the incisor, canine and premolar area and presence of two natural adjacent teeth
* no bone increasing procedures prior to and during dental implant,

Exclusion Criteria:

* history of a bleeding disorder or on anticoagulant therapy,
* immunocompromised state and debilitating disease,
* smoking and alcoholism,
* poor oral hygiene,
* diabetes.

Ages: 29 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Peri-implant Soft Tissue Thickness | Change from baseline soft tissue thickness at 3 months
  The measurement of soft tissue thickness at three points: occlusal part of the alveolar crest (OAC), midbuccal mucosa level (MBML), over 1 mm of mucogingival junction (MGJ1)]

SECONDARY OUTCOMES:
Keratinised Tissue Width (KTW) | Change from baseline keratinised tissue width at 3 months
  The measurement of the keratinised tissue width between the cover screw and the mucogingival junction.

CONTACTS AND LOCATIONS:
Overall Officials: Gülbahar Ustaoğlu, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Bolu Abant Izzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No